CLINICAL TRIAL: NCT02320513
Title: A Comparison of Physical Activity Levels With and Without Feedback Via Fitbit® Flex™ in Hemodialysis Patients
Acronym: IAM
Status: Completed | Type: Observational
Sponsor: Renal Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20141534
Record Dates: First submitted 2014-11-03; First posted 2014-12-19 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: End Stage Renal Disease
Keywords: Exercise
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group: Subjects will wear the activity monitoring device to track their activity between dialysis treatments, however, the feedback from the device will not be shared with them.
  Interventions: Other: Wearing activty monitoring device (Fitbit Flex); Device: Fitbit Flex
- Feedback Group: The feedback from the activity monitoring device will be shared with subjects at each visit.
  Interventions: Other: Wearing activty monitoring device (Fitbit Flex); Device: Fitbit Flex

INTERVENTIONS:
Other: Wearing activty monitoring device (Fitbit Flex)
Device: Fitbit Flex

SUMMARY:
This is a pilot study intended to gather data in order to inform future studies about the role of feedback as an incentive for increasing levels of physical activity which could improve health in hemodialysis patients.

DETAILED DESCRIPTION:
In prior studies that have analyzed physical activity in dialysis patients, three-dimensional accelerometers, physical performance tasks or self-reporting physical activity questionnaires have been used to measure levels of activity. This proposed study differs in that it will determine the effectiveness of providing "feedback" to dialysis patients using a fitness tracking bracelet. For the purpose of this study, the word 'feedback' is used to refer to the information provided to the subject that demonstrates the number of steps taken since the previous dialysis session as displayed by the Fitbit® application. This 'feedback' will allow subjects to be more aware of their overall physical activity on a quantitative level.

The study will seek to explore an association between feedback and physical activity. Improved physical activity could improve indicators of subjects' health status such as blood pressure, inflammatory markers, and pre-albumin levels, which will also be monitored and recorded.

While informing subjects quantitatively about their levels of physical activity could be a promising method to encourage them to be more active, it is unclear at this point if that strategy actually works. This is an important practical question though, because actually informing subjects on a regular basis about their activity level may pose substantial operative challenges and result in additional costs.

The importance of encouraging subjects to be more physically active should not be underestimated. Studying the physical activity of dialysis patients is important because it allows researchers to consider the long-term effects that may influence the subject's well-being. Johansen et al. showed that there was a direct relationship between the inactivity of dialysis patients and susceptibility to hypertension, diabetes, cardiovascular disease and even mortality. Additionally, the study demonstrated the importance of implementing programs to promote physical activity [1]. If feedback does indeed increase physical activity, then it will be substantially beneficial for this program to be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Receiving hemodialysis three times a week
* On hemodialysis for more than 3 months
* Between the ages of 18 and 75 years
* Able to walk without assistance or assistive devices
* Able to read and understand the English language

Exclusion Criteria:

* Patient already uses an activity tracker
* Unstable health: acute infections, congestive heart failure NYHA class 4 and/or unstable angina
* Hospitalization within the past 3 months for non-access related reasons
* Known allergies to nickel
* Unable to physically grip the handheld dynamometer in order to complete the Hand Grip Strength Test
* Cognitive impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Receiving hemodialysis three times a week
  * On hemodialysis for more than 3 months
  * Between the ages of 18 and 75 years
  * Able to walk without assistance or assistive devices
  * Able to read and understand the English language
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The effect of physical activity feedback on physical activity levels. | 5 weeks
  Physical activity level will be measured by the number of steps each subject takes. The number of steps each subject takes will be recorded and reported to those in one of the two groups. The study will evaluate whether a subject will begin to walk more steps once s/he is informed about the number of steps s/he is taking.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kotanko, MD, Principal Investigator — Renal Research Institute
Locations (1):
- Avantua Upper East Side Dialysis Center, New York, New York, United States